CLINICAL TRIAL: NCT02435849
Title: A Phase II, Single Arm, Multicenter Trial to Determine the Efficacy and Safety of CTL019 in Pediatric Patients With Relapsed and Refractory B-cell Acute Lymphoblastic Leukemia
Brief Title: Study of Efficacy and Safety of CTL019 in Pediatric ALL Patients
Acronym: ELIANA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTL019B2202; 2013-003205-25 (EudraCT Number)
Record Dates: First submitted 2015-04-16; First posted 2015-05-06 (Estimated); Results first posted 2021-11-22 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-12

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: Pediatric; ALL; Cell therapy; Lymphoblastic Leukemia; Acute; High Risk; Childhood; CTL019; tisagenlecleucel; Pediatric patients; r/r B-cell ALL; high risk B-cell ALL at first relapse; high risk B-cell ALL that relapsed < 6 months post allo-HSCT
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single dose of CTL019 (Experimental): Pediatric patients with relapsed or refractory B-cell ALL who were treated with single dose of tisagenlecleucel (CTL019).
  Interventions: Biological: CTL019

INTERVENTIONS:
Biological: CTL019 — Tisagenlecleucel was administered as a single iv infusion. Dose: 2.0 to 5.0x10^6 tisagenlecleucel per kg body weight (for patients ≤ 50 kg) or 1.0 to 2.5x10^8 tisagenlecleucel (for patients >50 kg).

SUMMARY:
This is a single arm, open-label, multi-center, phase II study to determine the efficacy and safety of CTL019 in pediatric patients with r/r B-cell ALL.

DETAILED DESCRIPTION:
This was a initially a one cohort, open-label, multi-center, phase II study to determine the efficacy and safety of CTL019 in pediatric patients with r/r B-cell ALL. This main cohort completed enrollment. Two new cohorts were added via an amendment, Cohort 1 for high risk B-cell ALL patients at first relapse, and Cohort 2 for feasibility and safety of CTL019 in high risk B-cell ALL in patients that relapsed <6 months post allo-HSCT. Due to lack of recruitment, Cohort 1 and Cohort 2 halted recruitment. This decision was not related to any safety issue.

The study had the following sequential phases: Screening, Pre-Treatment (Cell Product Preparation & Lymphodepleting Chemotherapy), Treatment and Primary Follow-up, Secondary Follow-up (if applicable) and Survival Follow-up. The total duration of the study is 5 years from CTL019 cell infusion.

Efficacy analyses were performed only on the Main Cohort (n=79) who were infused with tisagenlecleucel. However, the data on disposition and demographics presented in this section includes all patients enrolled to the study (98) and all infused patients (80) (Main Cohort + Cohort 1). No patients were enrolled in Cohort 2.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory pediatric B-cell ALL
2. Adequate organ function
3. For relapsed patients, documentation of CD19 tumor expression within 3 months of study entry.
4. Bone marrow with ≥ 5% lymphoblasts by morphologic assessment at screening.
5. Life expectancy > 12 weeks.
6. Karnofsky (age ≥16 years) or Lansky (age < 16 years) performance status ≥ 50 at screening
7. Signed written informed consent and assent forms
8. Must meet the institutional criteria to undergo leukapheresis or have an acceptable, store leukapheresis product
9. Must have an apheresis product of non-mobilized cells received and accepted by the manufacturing site.
10. Cohort 1 only:

    1. First relapse AND hypodiploid cytogenetics OR
    2. First relapse AND t(17;19) with defined TCF3-HLF fusion OR
    3. First relapse with any cytogenetics provided the relapse occurred ≤ 36 months of initial diagnosis AND MRD at end of reinduction therapy is ≥0.01% by flow cytometry (local assessment)

Exclusion Criteria

1. Isolated extra-medullary disease relapse
2. Patients with concomitant genetic syndrome: such as patients with Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome. Patients with Down Syndrome will not be excluded.
3. Patients with Burkitt's lymphoma/leukemia (i.e. patients with mature B-cell ALL, leukemia with B-cell [sIg positive and kappa or lambda restricted positivity] ALL, with FAB L3 morphology and /or a MYC translocation)
4. Prior malignancy, except carcinoma in situ of the skin or cervix treated with curative intent and with no evidence of active disease
5. Treatment with any prior gene therapy product
6. Has had treatment with any prior anti-CD19/anti-CD3 therapy, or any other anti-CD19 therapy
7. Active or latent hepatitis B or active hepatitis C (test within 8 weeks of screening), or any uncontrolled infection at screening
8. Human Immunodeficiency Virus (HIV) positive test within 8 weeks of screening
9. Presence of grade 2 to 4 acute or extensive chronic graft-versus-host disease (GVHD).
10. Active CNS involvement by malignancy, defined by CNS-3 per NCCN guidelines.
11. Patient has an investigational medicinal product within the last 30 days prior to screening.
12. Pregnant or nursing (lactating) women.
13. Women of child-bearing potential, defined as physiologically capable of becoming pregnant, unless they agree to use highly effective methods of contraception for at least 12 months after the CTL019 infusion and after CAR T-cells are no longer present by qPCR on two consecutive tests
14. Sexually active males must use a condom during intercourse at least 12 months after the CTL019 infusion after CAR T-cells are no longer present by qPCR on two consecutive tests

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (11):
  - Childrens Hospital Los Angeles SC CTL019, Los Angeles, California
  - Stanford Universtiy Medical Center SC - CTL019B2205J - B2206, Stanford, California
  - Children's Healthcare of Atlanta SC CTL019, Atlanta, Georgia
  - University of Michigan ., Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Children s Mercy Hospital SC - CTL019B2205J, Kansas City, Missouri
  - Duke Unversity Medical Center ., Durham, North Carolina
  - Oregon Health and Science University Doernbecher Children's Hosp., Portland, Oregon
  - The Childrens Hospital of Philadelphia CHOP, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center ., Dallas, Texas
  - University of Utah Clinical Trials Office SC - CTL019B2205J, Salt Lake City, Utah
- Novartis Investigative Site, Parkville, Victoria, Australia
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Ghent, Belgium
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (2):
  - Novartis Investigative Site, Paris, Cedex 10
  - Novartis Investigative Site, Paris
- Novartis Investigative Site, Frankfurt, Germany
- Novartis Investigative Site, Monza, MB, Italy
- Novartis Investigative Site, Kyoto, Japan
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Laetsch TW, Maude SL, Rives S, Hiramatsu H, Bittencourt H, Bader P, Baruchel A, Boyer M, De Moerloose B, Qayed M, Buechner J, Pulsipher MA, Myers GD, Stefanski HE, Martin PL, Nemecek E, Peters C, Yanik G, Khaw SL, Davis KL, Krueger J, Balduzzi A, Boissel N, Tiwari R, O'Donovan D, Grupp SA. Three-Year Update of Tisagenlecleucel in Pediatric and Young Adult Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia in the ELIANA Trial. J Clin Oncol. 2023 Mar 20;41(9):1664-1669. doi: 10.1200/JCO.22.00642. Epub 2022 Nov 18. PMID 36399695
- [Derived] Laetsch TW, Maude SL, Balduzzi A, Rives S, Bittencourt H, Boyer MW, Buechner J, De Moerloose B, Qayed M, Phillips CL, Pulsipher MA, Hiramatsu H, Tiwari R, Grupp SA. Tisagenlecleucel in pediatric and young adult patients with Down syndrome-associated relapsed/refractory acute lymphoblastic leukemia. Leukemia. 2022 Jun;36(6):1508-1515. doi: 10.1038/s41375-022-01550-z. Epub 2022 Apr 14. PMID 35422096
- [Derived] Thudium Mueller K, Grupp SA, Maude SL, Levine JE, Pulsipher MA, Boyer MW, August KJ, Myers GD, Tam CS, Jaeger U, Foley SR, Borchmann P, Schuster SJ, Waller EK, Awasthi R, Potthoff B, Warren A, Waldron ER, McBlane F, Chassot-Agostinho A, Laetsch TW. Tisagenlecleucel immunogenicity in relapsed/refractory acute lymphoblastic leukemia and diffuse large B-cell lymphoma. Blood Adv. 2021 Dec 14;5(23):4980-4991. doi: 10.1182/bloodadvances.2020003844. PMID 34432863
- [Derived] Levine JE, Grupp SA, Pulsipher MA, Dietz AC, Rives S, Myers GD, August KJ, Verneris MR, Buechner J, Laetsch TW, Bittencourt H, Baruchel A, Boyer MW, De Moerloose B, Qayed M, Davies SM, Phillips CL, Driscoll TA, Bader P, Schlis K, Wood PA, Mody R, Yi L, Leung M, Eldjerou LK, June CH, Maude SL. Pooled safety analysis of tisagenlecleucel in children and young adults with B cell acute lymphoblastic leukemia. J Immunother Cancer. 2021 Aug;9(8):e002287. doi: 10.1136/jitc-2020-002287. PMID 34353848
- [Derived] Buechner J, Grupp SA, Hiramatsu H, Teachey DT, Rives S, Laetsch TW, Yanik GA, Wood P, Awasthi R, Yi L, Chassot-Agostinho A, Eldjerou LK, De Moerloose B. Practical guidelines for monitoring and management of coagulopathy following tisagenlecleucel CAR T-cell therapy. Blood Adv. 2021 Jan 26;5(2):593-601. doi: 10.1182/bloodadvances.2020002757. PMID 33496754
- [Derived] Laetsch TW, Myers GD, Baruchel A, Dietz AC, Pulsipher MA, Bittencourt H, Buechner J, De Moerloose B, Davis KL, Nemecek E, Driscoll T, Mechinaud F, Boissel N, Rives S, Bader P, Peters C, Sabnis HS, Grupp SA, Yanik GA, Hiramatsu H, Stefanski HE, Rasouliyan L, Yi L, Shah S, Zhang J, Harris AC. Patient-reported quality of life after tisagenlecleucel infusion in children and young adults with relapsed or refractory B-cell acute lymphoblastic leukaemia: a global, single-arm, phase 2 trial. Lancet Oncol. 2019 Dec;20(12):1710-1718. doi: 10.1016/S1470-2045(19)30493-0. Epub 2019 Oct 9. PMID 31606419
- [Derived] Maude SL, Laetsch TW, Buechner J, Rives S, Boyer M, Bittencourt H, Bader P, Verneris MR, Stefanski HE, Myers GD, Qayed M, De Moerloose B, Hiramatsu H, Schlis K, Davis KL, Martin PL, Nemecek ER, Yanik GA, Peters C, Baruchel A, Boissel N, Mechinaud F, Balduzzi A, Krueger J, June CH, Levine BL, Wood P, Taran T, Leung M, Mueller KT, Zhang Y, Sen K, Lebwohl D, Pulsipher MA, Grupp SA. Tisagenlecleucel in Children and Young Adults with B-Cell Lymphoblastic Leukemia. N Engl J Med. 2018 Feb 1;378(5):439-448. doi: 10.1056/NEJMoa1709866. PMID 29385370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 98 patients met the eligibility criteria and apheresis was accepted by the manufacturing facility, 80 patients were infused in this study: 79 in the Main Cohort and 1 in Cohort 1. No patients were infused in Cohort 2. Patients could discontinue the trial after meeting the eligibility criteria and prior to tisagenlecleucel infusion.
Pre-assignment Details: This study was conducted in 11 countries with 23 sites.
Groups:
- Main Cohort: Single Dose of CTL019: Pediatric patients with relapsed or refractory B-cell ALL who were treated with single dose of tisagenlecleucel (CTL019).
- Cohort 1: Single Dose of CTL019: Pediatric B-ALL patients who are very high risk at first relapse.
Period: Overall Study
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Started (Started = Enrolled in All cohorts) | 79 | 1
Enrolled and Infused | 79 | 1
Discontinued Study Follow-up | 48 | 1
Completed (Completed = study follow-up completed) | 31 | 0
Not Completed | 48 | 1
Not completed — Death | 23 | 0
Not completed — Lack of Efficacy | 10 | 0
Not completed — New therapy for study indication | 8 | 0
Not completed — Subject/guardian decision | 5 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The Full analysis set comprised all patients who received infusion of tisagenlecleucel.
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019 | Total
Number analyzed (Participants) | 79 | 1 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12 (5.38) | 4 (NA) — NA: Standard deviation cannot be calculated for only 1 patient | 11.9 (5.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 0 | 34
  Male | 45 | 1 | 46
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 58 | 1 | 59
  Asian | 10 | 0 | 10
  Other | 11 | 0 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Remission Rate (ORR) as Determined by Independent Review Committee (IRC) Assessment.
Description: Evaluating the efficacy of tisagenlecleucel therapy from all manufacturing facilities as measured by overall remission rate (ORR) during the 3 months after tisagenlecleucel administration. ORR included complete response (CR) and CR with incomplete blood count recovery (CRi) as determined by an Independent Review Committee assessment. Per response criteria defined by National Comprehensive Cancer Network (NCCN), American Society of Hematology (ASH) and International Working Group (IWG) guidelines.
  CR is defined as:
  Bone marrow <5% blasts, Peripheral blood: Neutrophils >1.0 x 10^9/L, and Platelets >100 x 10^9/L and Circulating blasts <1% and No evidence of extramedullary disease, at least 7 days transfusion independency.
  CRi is defined as all the prior criteria being met, except that the following exists: Neutrophils ≤1.0 x 10^9/L, and/or Platelets ≤100 x 10^9/L, and/or Platelet and/or neutrophil transfusions ≤7 days before the date of the peripheral blood sample for disease assessment.
Time Frame: during the 3 months after tisagenlecleucel administration
Population: Full Analysis Set (FAS): The Full analysis set comprised all patients who received infusion of tisagenlecleucel in the Main Cohort.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 79 | 1
Percentage of participants | 82.3 [72.1 to 90.0] | 100.0 [NA to NA] — NA: Confidence Interval could not be calculated for only 1 participant.
Statistical Analysis 1: Comparison: Main Cohort: Single Dose of CTL019; Test type: Other — testing the null hypothesis that ORR within 3 months is less than or equal to 20%; p < .0001, Clopper-Pearson

2. Secondary Outcome: Percentage of Participants With Overall Remission Rate (ORR) as Per IRC From US Manufacturing Facilities in the Main Cohort Only (Key Secondary)
Description: These are the percentage of participants with ORR who achieved overall remission rate which includes complete response (CR) and CR with incomplete blood count recovery (CRi) as determined by IRC assessment after having been infused with tisagenlecleucel from US manufacturing facilities.
Time Frame: 3 months after tisagenlecleucel administration
Population: FAS: The Full analysis set comprised all patients who received infusion of tisagenlecleucel from US manufacturing facilities.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Cohort: Single Dose of CTL019
Number analyzed (Participants) | 67
Percentage of participants | 82.1 [70.8 to 90.4]

3. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) of CR or CRi With Minimal Residue Disease (MRD) Negative Bone Marrow From US Manufacturing Facility as Per IRC in the Main Cohort Only (Key Secondary)
Description: These are the percentage of participants who achieved Best Overall Response (BOR) of complete response (CR) or complete response with incomplete blood count recovery (CRi) with an MRD-negative bone marrow by central analysis using flow cytometry among participants who received tisagenlecleucel from US manufacturing facilities only, by IRC assessment.
Time Frame: 3 months after tisagenlecleucel administration
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Cohort: Single Dose of CTL019
Number analyzed (Participants) | 67
Percentage of participants | 82.1 [70.8 to 90.4]
Statistical Analysis 1: Comparison: Main Cohort: Single Dose of CTL019; Test type: Other — testing the null hypothesis that ORR with MRD negative within 3 months is less than or equal to 15%; p < .0001, Clopper-Pearson

4. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) of CR or CRi With MRD Negative Bone Marrow by Flow Cytometry From All Manufacturing Facilities as Per IRC in the Main Cohort Only (Key Secondary)
Description: These are the percentage of participants who achieved Best Overall Response (BOR) of CR or CRi with an MRD-negative bone marrow by central analysis using flow cytometry among participants who received tisagenlecleucel from all manufacturing facilities by IRC assessment. MRD negative = MRD% < 0.01%
Time Frame: 3 months after tisagenlecleucel administration
Population: FAS: The Full analysis set comprised all patients who received infusion of tisagenlecleucel from all manufacturing facilities.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Cohort: Single Dose of CTL019
Number analyzed (Participants) | 79
Percentage of participants | 81.0 [70.6 to 89.0]
Statistical Analysis 1: Comparison: Main Cohort: Single Dose of CTL019; Test type: Other — testing the null hypothesis that ORR with MRD negative within 3 months is less than or equal to 15%; p < .0001, Clopper-Pearson

5. Secondary Outcome: Percentage of Participants Who Achieved CR or CRi Without Hematopoietic Stem Cell Transplantation (HSCT)
Description: These are the participants who achieved CR or CRi without HSCT between tisagenlecleucel (CTL019) infusion and Month 6 response assessment.
Time Frame: 6 months after tisagenlecleucel administration
Population: FAS: The Full analysis set comprised all patients who received infusion of tisagenlecleucel.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 79 | 1
Percentage of participants | 60.8 [49.1 to 71.6] | 100.0 [NA to NA] — NA: Confidence Interval could not be calculated for only 1 participant.

6. Secondary Outcome: Percentage of Participants Who Achieved CR or CRi and Then Proceeded to Hematopoietic Stem Cell Transplantation (HSCT) While in Remission Prior to Month 6 Resoonse
Description: These are the participants who achieved CR or CRi and then proceeded to HSCT while in remission prior to Month 6 response assessment
Time Frame: 6 months
Population: FAS: The Full analysis set comprised all patients who received infusion of tisagenlecleucel.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 79 | 1
Percentage of Participants | 7.6 [2.8 to 15.8] | 0.0 [NA to NA] — NA: Confidence Interval could not be calculated for only 1 participant.

7. Secondary Outcome: Number of Participants Who Proceeded to Hematopoietic Stem Cell Transplantation (HSCT) After Tisagenlecleucel (CTL019) Infusion
Description: These are the participants who achieved CR or CRi and then proceeded to SCT after being infused by tisagenlecleucel.
Time Frame: up to 6 months
Population: FAS: The Full analysis set comprised all patients who received infusion of tisagenlecleucel.
Measure: Number; unit: Participants
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 79 | 1
Participants | 18 | 0

8. Secondary Outcome: Duration of Remission (DOR)
Description: DOR is the time from achievement of CR or CRi at any time post-infusion, whichever occurs first, to relapse or death.
Time Frame: 60 months
Population: FAS: The Full analysis set comprised all patients who received infusion of tisagenlecleucel and who achieved CR or CRi.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 66 | 1
months | 46.8 [17.8 to NA] — NA: more than 50% were either censored or in remission at time of analysis. | NA [NA to NA] — NA: The patient did not relapse at the time of discontinuation.

9. Secondary Outcome: Site of Involvement of Subsequent Relapse
Description: Anatomical location of relapse in participants who achieved prior CR/CRi subsequent to tisagenlecleucel infusion.
Time Frame: 60 months
Population: FAS: The Full analysis set comprised all patients who received infusion of tisagenlecleucel and who achieved CR or CRi. Achieving CR or CRi" requireb confirmation but for this analysis, all patients with one CR/CRi, regardless of confirmation were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 71 | 0
Participants
  BM and/or blood relapse | 23 |
  Extramedullary only | 2 |
  Unknown | 4 |

10. Secondary Outcome: Relapse-free Survival Per IRC Assessment
Description: RFS is the time from achievement of CR or CRi at any time post-infusion, whichever occurs first, to relapse or death due to any cause during CR or CRi.
Time Frame: 60 months
Population: FAS: The Full analysis set comprised all patients who received infusion of tisagenlecleucel.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 66 | 1
months | 46.8 [17.8 to NA] — NA: more than 50% were either censored or in remission at time of analysis. | NA [NA to NA] — NA: The patient did not relapse at the time of discontinuation.

11. Secondary Outcome: Event-free Survival Per IRC Assessment
Description: EFS is the time from date of tisagenlecleucel infusion to the earliest of death, relapse or treatment failure.
Time Frame: 60 months
Population: FAS: The Full analysis set comprised all patients who received infusion of tisagenlecleucel
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 79 | 1
months | 23.7 [9.2 to NA] — NA: more than 50% were either censored or without failure event at time of analysis. | NA [NA to NA] — NA: The patient did not have an EFS event at the time of discontinuation.

12. Secondary Outcome: Overall Survival (OS)
Description: OS, is the time from date of tisagenlecleucel infusion to the date of death due to any reason.
Time Frame: 60 months
Population: FAS: The Full analysis set comprised all patients who received infusion of tisagenlecleucel
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 79 | 1
months | NA [45.6 to NA] — NA: median was not reached, simply because more than 50% of patients remained alive at end of study, or data was otherwise censored. | NA [NA to NA] — NA: The patient was still alive at the time of discontinuation.

13. Secondary Outcome: Percentage of Participants Attaining CR or CRi at Day 28 +/- 4 Days Post Tisagenlecleucel (CTL019) Infusion by IRC Assessment
Description: These are participants who had a day 28 response (CR or CRi response) by IRC assessment.
Time Frame: 1 month
Population: FAS: The Full analysis set comprised all patients who received infusion of tisagenlecleucel.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 79 | 1
Percentage of participants | 78.5 [67.8 to 86.9] | 100 [NA to NA] — NA: Confidence Interval could not be calculated for only 1 participant.

14. Secondary Outcome: Response as a Function of Baseline Tumor Burden (Tumor Load) in Main Cohort Only
Description: Percentage of participants who achieved BOR of CR or CRi by flow cytometry as a function of baseline bone marrow tumor burden.
Time Frame: 3 months
Population: FAS: The Full analysis set comprised all patients who received infusion of tisagenlecleucel with a baseline tumor burden assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 79 | 1
Percentage of participants
  Baseline bone marrow tumor burden: Low (<50%): number analyzed (Participants) | 25 | 1
  Baseline bone marrow tumor burden: Low (<50%) | 96.0 [79.6 to 99.9] | 100.0 [NA to NA] — NA: 95% CI could not be calculated as there was only 1 participant who had low baseline tumor burden
  Baseline bone marrow tumor burden: High (>=50%): number analyzed (Participants) | 54 | 0
  Baseline bone marrow tumor burden: High (>=50%) | 75.9 [62.4 to 86.5] |

15. Secondary Outcome: Bone Marrow MRD Status by Flow Cytometry Per IRC Assessment
Description: Percentage of participants who achieved CR or CRi response with bone marrow MRD negative (MRD < 0.01%) after tisagenlecleucel infusion by flow cytometry.
Time Frame: 28 days
Population: FAS: The Full analysis set comprised all patients who received infusion of tisagenlecleucel
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 79 | 1
Percentage of participants | 75.9 [65.0 to 84.9] | 100.0 [NA to NA] — NA: Confidence Interval could not be calculated for only1 participant.

16. Secondary Outcome: Tisagenlecleucel Transgene Levels by qPCR in Peripheral Blood by Day 28 Response by Independent Review Committee (IRC) Assessment
Description: This is the summary of cellular kinetic concentrations for Tisagenlecleucel (CTL019) transgene levels by qPCR in peripheral blood.
Time Frame: Month 60
Population: PAS: The PAS consisted of patients in the FAS who had at least one sample providing evaluable cellular kinetic data for tisagenlecleucel. Analysis of this particular outcome included a subset of PAS who had evaluation data of the parameter at the specific timepoint. Therefore, no participants in Cohort 1 had at least one blood sample providing evaluable cellular kinetic data for tisagenlecleucel at tis time point, so no data was collected for Cohort 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/ug DNA
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 20 | 0
copies/ug DNA | 207 (95.5) |

17. Secondary Outcome: Tisagenlecleucel Transgene Levels by qPCR in Bone Marrow by Day 28 Response by IRC Assessment
Description: This is the summary of cellular kinetic concentrations for Tisagenlecleucel (CTL019) transgene levels by qPCR in bone marrow.
Time Frame: Month 6
Population: PAS: The PAS consisted of patients in the FAS who had at least one sample providing evaluable cellular kinetic data for tisagenlecleucel parameter under investigation. Analysis of this particular outcome included a subset of PAS who had evaluation data of the parameter at the specific timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/ug DNA
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 39 | 1
copies/ug DNA | 210 (138.1) | NA (NA) — NA: Geometric mean/Geometric Coefficient of Variation could not be calculated for only 1 participant

18. Secondary Outcome: Expression of Tisagenlecleucel (CTL019) Detected by Flow Cytometry in Peripheral Blood by Day 28 Disease Response Per IRC Assessment
Description: This is the summary cellular kinetic concentrations for CTL019 by flow cytometry in peripheral blood. It evaluated the persistence of transduced CTL019 cells post-infusion. Observation was up to Month 60 for peripheral blood.
Time Frame: Month 60
Population: PAS: The PAS consisted of patients in the FAS who had at least one sample providing evaluable cellular kinetic data for tisagenlecleucel parameter under investigation. Analysis of this particular outcome included a subset of PAS who had evaluation data of the parameter at the specific timepoint. Therefore, no participants in Cohort 1 had at least one blood sample providing evaluable cellular kinetic data for tisagenlecleucel at tis time point, so no data was collected for Cohort 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of CD3+/CTL019+ cells
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 17 | 0
Percentage of CD3+/CTL019+ cells | 0.253 (67.4) |

19. Secondary Outcome: Expression of Tisagenlecleucel (CTL019) Detected by Flow Cytometry in Bone Marrow by Day 28 Response by IRC Assessment
Description: This is the summary cellular kinetic concentrations for CTL019 by flow cytometry. It evaluated the persistence of transduced CTL019 cells post-infusion. Observation was up to Month 6 for bone marrow.
Time Frame: Month 6
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of CD3+/CTL019+ cells
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 49 | 1
Percentage of CD3+/CTL019+ cells | 0.519 (185.8) | 0.1 (NA) — NA: Geo-CV could not be calculated for only 1 participant.

20. Secondary Outcome: Pharmacokinetics (PK) Parameter: Cmax by qPCR in Peripheral Blood, by Day 28 Disease Response by IRC
Description: Cmax is the maximum (peak) observed in peripheral blood drug concentration after single dose administration reported by CR/CRi, no response (NR), Unknown and by All participants. D28 refers to the timepoint for definition of responder populations, whereas M60 is the actual timepoint for endpoint assessment. The reported Cmax is the summary of maximum level observed based on the data from each patient and based on all the data that's been collected for up to 60 months in a patient.
Time Frame: 60 months
Population: PAS: The PAS consisted of patients in the FAS who had at least one sample providing evaluable cellular kinetic data for tisagenlecleucel.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/ug
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 75 | 1
copies/ug
  CR/CRi: number analyzed (Participants) | 62 | 1
  CR/CRi | 37200 (154.2) | 2690 (NA) — NA: Geo-CV could not be calculated for 1 participant.
  NR: number analyzed (Participants) | 5 | 0
  NR | 31700 (87.4) |
  Unknown: number analyzed (Participants) | 8 | 0
  Unknown | 67700 (132.5) |
  All Participants | 39200 (148.8) | 2690 (NA) — NA: Geo-CV could not be calculated for 1 participant.

21. Secondary Outcome: Pharmacokinetics (PK) Parameter: Tmax by qPCR in Peripheral Blood, by Day 28 Disease Response by IRC
Description: Tmax is the time to reach maximum (peak) peripheral blood drug concentration after single dose administration (days)", reported by CR/CRi, no response (NR), Unknown and by All participants. D28 refers to the timepoint for definition of responder populations, whereas M60 is the actual timepoint for endpoint assessment. The time frame of 60 months refers to the duration for which the data were reviewed to identify the time of Cmax for this measure.
Time Frame: 60 months
Population: as for outcome 20
Measure: Median (Full Range); unit: days
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 75 | 1
days
  CR/CRi: number analyzed (Participants) | 62 | 1
  CR/CRi | 9.87 [5.70 to 27.8] | 8.55 [8.55 to 8.55]
  NR: number analyzed (Participants) | 5 | 0
  NR | 20.9 [12.6 to 62.7] |
  Unknown: number analyzed (Participants) | 8 | 0
  Unknown | 13.4 [8.73 to 19.9] |
  All Participants | 9.98 [5.70 to 62.7] | 8.55 [8.55 to 8.55]

22. Secondary Outcome: Pharmacokinetics (PK) Parameter: AUCs by qPCR in Peripheral Blood, by Day 28 Disease Response by IRC
Description: AUC (area under curve) from day of infusion to day 28 or other disease assessment days, in peripheral blood (% or copies/μg x days), reported by CR/CRi, no response (NR), Unknown and by All participants. D28 refers to the timepoint for definition of responder populations, whereas 84 days is the actual timepoint for endpoint assessment. : AUC is defined based on the time window i.e., AUC from 0 to 84 days after infusion. Therefore, the time frame specifies the maximum time for up to which the data are used for estimation of AUC (84 days for AUC84d).
Time Frame: 0 to 84 days after infusion
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/ug*days
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 75 | 1
copies/ug*days
  AUC0-28d: CR/CRi: number analyzed (Participants) | 62 | 1
  AUC0-28d: CR/CRi | 310000 (192.2) | 31500 (NA) — NA: Geo-CV could not be calculated for 1 participant.
  AUC0-28d: NR: number analyzed (Participants) | 5 | 0
  AUC0-28d: NR | 301000 (116.9) |
  AUC0-28d: Unknown: number analyzed (Participants) | 8 | 0
  AUC0-28d: Unknown | 768000 (177.4) |
  AUC0-28d: All Participants | 341000 (190.9) | 31500 (NA) — NA: Geo-CV could not be calculated for 1 participant.
  AUC 0-84d: CR/CRi: number analyzed (Participants) | 56 | 1
  AUC 0-84d: CR/CRi | 462000 (230.1) | 74700 (NA) — NA: Geo-CV could not be calculated for 1 participant.
  AUC 0-84d: NR: number analyzed (Participants) | 3 | 0
  AUC 0-84d: NR | 1130000 (75.5) |
  AUC 0-84d: Unknown: number analyzed (Participants) | 7 | 0
  AUC 0-84d: Unknown | 984000 (202.4) |
  AUC 0-84d: All Participants: number analyzed (Participants) | 66 | 1
  AUC 0-84d: All Participants | 521000 (225.3) | 74700 (NA) — NA: Geo-CV could not be calculated for 1 participant.

23. Secondary Outcome: Persistence of Tisagenlecleucel (CTL019) in Blood, Bone Marrow and CSF if Available, by qPCR, by Day 28 Response by IRC
Description: Persistence is defined as the time corresponding to last quantifiable transgene level in peripheral blood (Tlast), reported by CR/CRi, no response (NR), Unknown and by All participants. D28 refers to the timepoint for definition of responder populations, whereas M60 is the actual timepoint for endpoint assessment.
Time Frame: 60 months
Population: as for outcome 20
Measure: Median (Full Range); unit: days
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 76 | 1
days
  Tlast CR/CRi: number analyzed (Participants) | 62 | 1
  Tlast CR/CRi | 232 [19.8 to 1860] | 89.7 [89.7 to 89.7]
  Tlast NR: number analyzed (Participants) | 6 | 0
  Tlast NR | 48.5 [13.9 to 888] |
  Tlast Unknown: number analyzed (Participants) | 8 | 0
  Tlast Unknown | 220 [64.0 to 1460] |
  Tlast All Participants | 179 [13.9 to 1860] | 89.7 [89.7 to 89.7]

24. Secondary Outcome: Prevalence and Incidence of Immunogenicity to Tisagenlecleucel (CTL019)
Description: This is defined as the percentage of participants who tested positive for anti-mCAR19 antibodies at any time post-baseline, reported by CR/CRi, no response (NR), Unknown and by All participants. .
Time Frame: At any time post-baseline, up to a max. of 60 months
Population: Safety Set: The Safety set comprised all patients who received tisagenlecleucel infusion in the Main Cohort. No participants in Cohort 1 had immunogenicity data providing evaluable cellular kinetic data for tisagenlecleucel at this time point, so no data was collected for Cohort 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 79 | 0
Participants
  CR/CRi positive: number analyzed (Participants) | 62 | 0
  CR/CRi positive | 61 |
  NR positive: number analyzed (Participants) | 6 | 0
  NR positive | 6 |
  Unknown positive: number analyzed (Participants) | 11 | 0
  Unknown positive | 11 |
  All Patients positive | 78 |

25. Secondary Outcome: Effects of CTL019 Therapy on Patient Reported Outcomes as Measured by PedsQL Questionnaire
Description: The PedsQL questionnaire was for patients ≥ 8-years-old who achieved BOR as CR or CRi within 3 months and the questionnaire was on emotional, social, school, physical, and psychosocial health. Scores are transformed on a scale from 0 to 100, with the sum of all the items over the number of items answered on all the scales. The total scale score is the averaged value of scores of subscales, which means for each subscale and the total scale, the allowed ranges are 0-100. Higher scores on the PedsQL questionnaire for these subscales indicate consistent improvement of health-related quality of life (HRQol).
Time Frame: Month 3, M6, M12, M24, M60
Population: FAS: the Full analysis set comprised all patients who received infusion of tisagenlecleucel and who had evaluable results at the measured time points. This analysis included a subset of FAS who had any data of the particular questionnaire at the specific timepoint. Therefore, no participants in Cohort 1 had questionnaire data for tisagenlecleucel at the measured time points, so no data was collected for Cohort 1.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 39 | 0
Scores on a scale
  M3 change from baseline - Emotional | 14.5 (17.98) |
  M6 change from baseline - Emotional: number analyzed (Participants) | 37 | 0
  M6 change from baseline - Emotional | 15.9 (18.96) |
  M12 change from baseline - Emotional: number analyzed (Participants) | 23 | 0
  M12 change from baseline - Emotional | 24.6 (23.74) |
  M24 change from baseline - Emotional: number analyzed (Participants) | 20 | 0
  M24 change from baseline - Emotional | 27.02 (21.85) |
  M60 change from baseline - Emotional: number analyzed (Participants) | 14 | 0
  M60 change from baseline - Emotional | 21.4 (24.53) |
  M3 change from baseline - Social | 7.6 (13.90) |
  M6 change from baseline - Social: number analyzed (Participants) | 37 | 0
  M6 change from baseline - Social | 8.4 (17.04) |
  M12 change from baseline - Social: number analyzed (Participants) | 23 | 0
  M12 change from baseline - Social | 14.8 (16.68) |
  M24 change from baseline - Social: number analyzed (Participants) | 20 | 0
  M24 change from baseline - Social | 17.3 (15.85) |
  M60 change from baseline - Social: number analyzed (Participants) | 14 | 0
  M60 change from baseline - Social | 17.9 (14.77) |
  M3 change from baseline - School: number analyzed (Participants) | 30 | 0
  M3 change from baseline - School | 8.9 (14.35) |
  M6 change from baseline - School: number analyzed (Participants) | 29 | 0
  M6 change from baseline - School | 10.0 (16.58) |
  M12 change from baseline - School: number analyzed (Participants) | 20 | 0
  M12 change from baseline - School | 19.0 (19.97) |
  M24 change from baseline - School: number analyzed (Participants) | 18 | 0
  M24 change from baseline - School | 13.9 (23.98) |
  M60 change from baseline - School: number analyzed (Participants) | 13 | 0
  M60 change from baseline - School | 17.7 (24.46) |
  M3 change from baseline - Physical | 17.5 (18.36) |
  M6 change from baseline - Physical: number analyzed (Participants) | 37 | 0
  M6 change from baseline - Physical | 21.6 (25.81) |
  M12 change from baseline - Physical: number analyzed (Participants) | 23 | 0
  M12 change from baseline - Physical | 31.1 (28.57) |
  M24 change from baseline - Physical: number analyzed (Participants) | 20 | 0
  M24 change from baseline - Physical | 37.4 (25.12) |
  M60 change from baseline - Physical: number analyzed (Participants) | 14 | 0
  M60 change from baseline - Physical | 37.1 (24.90) |
  M3 change from baseline - Psychosocial health | 10.4 (12.38) |
  M6 change from baseline - Psychosocial health: number analyzed (Participants) | 37 | 0
  M6 change from baseline - Psychosocial health | 11.0 (14.08) |
  M12 change from baseline - Psychosocial health: number analyzed (Participants) | 23 | 0
  M12 change from baseline - Psychosocial health | 19.8 (16.80) |
  M24 change from baseline - Psychosocial health: number analyzed (Participants) | 20 | 0
  M24 change from baseline - Psychosocial health | 20.1 (16.34) |
  M60 change from baseline - Psychosocial health: number analyzed (Participants) | 14 | 0
  M60 change from baseline - Psychosocial health | 18.9 (15.15) |
  M3 change from baseline - Total score | 13.0 (13.28) |
  M6 change from baseline - Total score: number analyzed (Participants) | 37 | 0
  M6 change from baseline - Total score | 14.8 (17.00) |
  M12 change from baseline - Total score: number analyzed (Participants) | 23 | 0
  M12 change from baseline - Total score | 2.8 (19.56) |
  M24 change from baseline - Total score: number analyzed (Participants) | 20 | 0
  M24 change from baseline - Total score | 26.2 (16.70) |
  M60 change from baseline - Total score: number analyzed (Participants) | 14 | 0
  M60 change from baseline - Total score | 25.3 (15.45) |

26. Secondary Outcome: Effects of CTL019 Therapy on Patient Reported Outcomes as Measured by EQ-5D Questionnaire
Description: Results from the EQ-5D questionnaire is for number of participants who achieved CR or CRi at month 60. The EQ-5D descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain & discomfort, anxiety & depression. Respondents are asked to choose the statement in each dimension that best describes their health status on the day surveyed. Their responses are coded as a number (1, 2, or 3) that corresponds to the respective level of severity: 1 indicates no problems, 2 some problems, and 3 severe problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the 5 dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the 5 dimensions can be combined into a 5-digit number that describes the patient's health state. The scores are then normalized to a value from 0-100 where higher scores = better HRQOL & fewer problems or symptoms.
Time Frame: Month 60
Population: FAS: The Full analysis set comprised all patients who received infusion of tisagenlecleucel and who had evaluable results at the measured time points. This analysis included a subset of FAS who had any data of the particular questionnaire at the measured timepoints. Therefore, no participants in Cohort 1 had questionnaire data for tisagenlecleucel at the measured time points, so no data was collected for Cohort 1.
Measure: Number; unit: Participants
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 16 | 0
Participants
  M60: Mobility - No problems | 15 |
  M60: Mobility - Some problems | 1 |
  M60: Mobility - Severe problems | 0 |
  M60: Self-care - No problems | 16 |
  M60: Self-care - Some problems | 0 |
  M60: Self-care - Severe problems | 0 |
  M60: Usual activities - No problems | 15 |
  M60: Usual activities - Some problems | 0 |
  M60: Usual activities - Severe problems | 1 |
  M60: Pain/discomfort - No problems | 14 |
  M60: Pain/discomfort - Some problems | 2 |
  M60: Pain/discomfort - Severe problems | 0 |
  M60: Anxiety/depression - No problems | 12 |
  M60: Anxiety/depression - Some problems | 4 |
  M60: Anxiety/depression - Severe problems | 0 |

27. Secondary Outcome: Develop a Score Utilizing Clinical and Biomarker Data and Assess Its Ability for Early Prediction of Cytokine Release Syndrome (CRS)
Description: Derivation of a score to predict cytokine release syndrome. Considering the complexity and challenges of building a scoring system based on limited data from the trial, this analysis was not performed.
Time Frame: 3 months
Population: This objective was not associated with any data collection from participants. The original plan was to mathematically derive a score from other endpoints measures (e.g., a score combing age, value of CRP, Ferritin, Interferon gamma, etc.). Those potential biomarkers were used to derive the scores that are already reported in other tables. None of the biomarkers analyzed proved to be prognostic for the onset or severity of CRS, hence finally no score was derived and no data for this objective.
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Frequent Monitoring of Concentrations of Soluble Immune Factors in Blood (C Reactive Protein & Ferritin)
Description: Profile of soluble immune factors of key inflammatory markers and cytokine parameters in blood by maximum CRS grade that may be key to cytokine release syndrome (CRS).
Time Frame: Maximum post-baseline (approx. 60 months)
Population: Safety Set: The Safety set comprised all patients who received tisagenlecleucel infusion with evaluable data. This analysis included a subset of Safety set who had any data of the particular biomarker at the specific timepoint. Therefore, no participants in Cohort 1 had biomarker data at this time point, so no data was collected for Cohort 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: fold-change from baseline
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 21 | 0
fold-change from baseline
  C Reactive Protein: Fold-change from BL Grade 4 CRS | 9.33 (303.9) |
  Ferritin: Fold-change from BL Grade 4 CRS | 36.62 (164.6) |

29. Secondary Outcome: Frequent Monitoring of Concentrations of Soluble Immune Factors in Blood (All Other Inflammatory Markers)
Description: as for outcome 28
Time Frame: Maximum post-baseline (approx. 60 months)
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: fold-change from baseline
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 21 | 0
fold-change from baseline
  Interferon gamma: Fold-change from BL Grade 4 CRS | 2745.92 (1186.3) |
  Interleukin 10: Fold-change from BL Grade 4 CRS | 179.49 (966.7) |
  Interleukin 12p70: Fold-change from BL Grade 4 CRS | 93.50 (261.0) |
  Interleukin 13: Fold-change from BL Grade 4 CRS | 49.21 (124.0) |
  Interleukin 1 beta: Fold-change from BL Grade 4 CRS | 16.75 (127.7) |
  Interleukin 2: Fold-change from BL Grade 4 CRS | 337.86 (161.1) |
  Interleukin 4: Fold-change from BL Grade 4 CRS | 170.21 (163.3) |
  Interleukin 6: Fold-change from BL Grade 4 CRS | 1435.85 (221.6) |
  Interleukin 8: Fold-change from BL Grade 4 CRS | 139.40 (246.9) |
  Tumor necrosis factor alpha: Fold-change from BL Grade 4 CRS | 27.13 (223.7) |

30. Secondary Outcome: Percentage Change From Baseline of Levels of B and T Cells (Blood and Bone Marrow) Prior to and Following CTL019 Infusion
Description: Levels of B and T cells (blood and bone marrow) prior to and following CTL019 infusion for safety monitoring
Time Frame: Month 3, Month 12, Maximum post-baseline (approx. 60 months)
Population: Safety Set: The Safety set comprised all patients who received tisagenlecleucel infusion.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 79 | 1
percentage change from baseline
  M3: % change from BL - (B cell) CR/CRi: number analyzed (Participants) | 57 | 1
  M3: % change from BL - (B cell) CR/CRi | -25.37 (31.693) | -0.51 (NA) — NA: not enough participants to analyze the Standard Deviation.
  M3: % change from BL - (B cell) NR: number analyzed (Participants) | 3 | 0
  M3: % change from BL - (B cell) NR | -37.93 (35.882) |
  M3: % change from BL - (B cell) Unknown: number analyzed (Participants) | 8 | 0
  M3: % change from BL - (B cell) Unknown | -11.01 (6.649) |
  M3: % change from BL - (B cell) All participants: number analyzed (Participants) | 68 | 1
  M3: % change from BL - (B cell) All participants | -24.23 (30.215) | -0.51 (NA) — NA: not enough participants to analyze the Standard Deviation.
  M12: % change from BL - (B cell) CR/CRi: number analyzed (Participants) | 34 | 0
  M12: % change from BL - (B cell) CR/CRi | -18.55 (27.144) |
  M12: % change from BL - (B cell) NR: number analyzed (Participants) | 1 | 0
  M12: % change from BL - (B cell) NR | -55.21 (NA) — NA: not enough participants to analyze the Standard Deviation. |
  M12: % change from BL - (B cell) Unknown: number analyzed (Participants) | 3 | 0
  M12: % change from BL - (B cell) Unknown | -12.04 (5.995) |
  M12 % change from BL -: (B cell) All Participants: number analyzed (Participants) | 38 | 0
  M12 % change from BL -: (B cell) All Participants | -19.00 (26.432) |
  Maximum post-BL: (B cell) CR/CRi: number analyzed (Participants) | 49 | 1
  Maximum post-BL: (B cell) CR/CRi | -21.25 (37.618) | 6.06 (NA) — NA: not enough participants to analyze the Standard Deviation.
  Maximum post-BL: (B cell) NR: number analyzed (Participants) | 5 | 0
  Maximum post-BL: (B cell) NR | 2.10 (66.398) |
  Maximum post-BL: (B cell) Unknown: number analyzed (Participants) | 8 | 0
  Maximum post-BL: (B cell) Unknown | 7.98 (29.536) |
  Maximum post-BL: (B cell) All participants: number analyzed (Participants) | 62 | 1
  Maximum post-BL: (B cell) All participants | -15.60 (40.336) | 6.06 (NA) — NA: not enough participants to analyze the Standard Deviation.
  M3: % change from BL - (T cell) All participants: number analyzed (Participants) | 67 | 0
  M3: % change from BL - (T cell) All participants | -11.91 (32.333) |
  M12: % change from BL - (T cell) All participants: number analyzed (Participants) | 38 | 0
  M12: % change from BL - (T cell) All participants | -1.68 (36.228) |
  Maximum post-BL: (T cell) All participants: number analyzed (Participants) | 41 | 0
  Maximum post-BL: (T cell) All participants | 34.12 (29.450) |

31. Secondary Outcome: Percentage of Participants With Overall Remission Rate (ORR) - From Fraunhofer Institute Manufacturing Facility
Description: These are the percentage of participants with ORR who achieved overall remission rate which includes complete response (CR) and CR with incomplete blood count recovery (CRi) as determined by IRC assessment after having been infused with tisagenlecleucel from Fraunhofer Institute manufacturing facility.
Time Frame: 60 months
Population: FAS: The Full analysis set comprised all patients who received infusion of tisagenlecleucel from Fraunhofer Institue Manufacturing Facility. Participants in Cohort 1 were from the Fraunhofer Institute manufacturing facility and not the US where the data was collected from, so no data was collected for this Cohort.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 12 | 0
Percentage of participants | 83.3 [51.6 to 97.9] |

32. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) of CR or CRi With Minimal Residue Disease (MRD) Negative Bone Marrow From Fraunhofer Institute Manufacturing Facility as Per IRC
Description: These are the percentage of participants who achieved Best Overall Response (BOR) of CR or CRi with an MRD-negative bone marrow by central analysis using flow cytometry among participants who received tisagenlecleucel from Fraunhofer Institute manufacturing facilities only, by IRC assessment.
Time Frame: 3 months
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 12 | 0
Percentage of participants | 75.0 [42.8 to 94.5] |

33. Secondary Outcome: Tisagenlecleucel Transgene Levels by qPCR in Peripheral Blood - Tisagenlecleucel Manufactured From Fraunhofer Institute
Description: This is the summary of cellular kinetic concentrations for Tisagenlecleucel (CTL019) transgene levels by qPCR, by disease response in blood by IRC assessment. The assessment of the efficacy, safety and in vivo cellular pharmacokinetics are for patients infused with tisagenlecleucel manufactured by Fraunhofer Institute.
Time Frame: Month 60
Population: PAS: The PAS consisted of patients in the FAS who had at least one sample providing evaluable cellular kinetic data for tisagenlecleucel from Fraunhofer Institue Manufacturing Facility. Participants in Cohort 1 were from the Fraunhofer Institute manufacturing facility and not the US where the data was collected from, so no data was collected for this Cohort.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: copies/ug
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 10 | 0
copies/ug | 42800 (117.7) |

34. Secondary Outcome: Tisagenlecleucel Transgene Levels by qPCR in Bone Marrow - Tisagenlecleucel Manufactured From Fraunhofer Institute
Description: This is the summary of cellular kinetic concentrations for Tisagenlecleucel (CTL019) transgene levels by qPCR, by disease response in bone marrow by IRC assessment. The assessment of the efficacy, safety and in vivo cellular pharmacokinetics are for patients infused with tisagenlecleucel manufactured by Fraunhofer Institute.
Time Frame: Month 3
Population: PAS: The PAS consisted of patients in the FAS who had at least one sample providing evaluable cellular kinetic data for tisagenlecleucel. Participants in Cohort 1 were from the Fraunhofer Institute manufacturing facility and not the US where the data was collected from, so no data was collected for this Cohort.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: copies/ug
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 7 | 0
copies/ug | 855 (792.6) |

35. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths, which include post-treatment survival follow-up deaths, were collected during the post-infusion period (starting at the day of first infusion) until the end of the study, approx. 60 months.
  All deaths refers to the sum of on-treatment deaths and post-treatment survival follow-up deaths up to approx. 60 months.
Time Frame: On-treatment deaths: Up to 60 months; Post-treatment survival follow-up deaths: Up to approx. 60 months
Population: Clinical Database Population: all infused participants in the Main cohort
Measure: Number; unit: Participants
Arm/Group | Main Cohort: Single Dose of CTL019 | Cohort 1: Single Dose of CTL019
Number analyzed (Participants) | 79 | 1
Participants
  On-treatment deaths include post-treatment survival follow-up deaths | 33 | 0
  All deaths | 33 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) timeframe: AEs were collected during the post-infusion period (starting at the day of 1st infusion until the end of the study), up to maximum duration of 60 months for each patient. Deaths were collected at all points post-treatment (including post-treatment survival follow-up period) until the patient completed the study duration (60 months) or further safety follow-up under the study protocol. Therefore on-treatment deaths include post-treatment survival follow-up deaths.
Description: AE description: Any sign or symptom that occurs during the post-infusion period (starting at the day of first infusion of CTL019 until the end of the study) and safety follow-up. Deaths in the post treatment survival follow-up are not considered Adverse Events while still included in the All-Cause Mortality table.
Groups:
- Main Cohort (On-treatment + Post-treatment Survival Follow-up Deaths): Single dose of CTL019Edit Pediatric patients with relapsed or refractory B-cell ALL who were treated with single dose of tisagenlecleucel (CTL019).
- Cohort 1 (On-treatment + Post-treatment Survival Follow-up Deaths): Single dose of CTL019Edit Pediatric B-ALL patients who are very high risk at first relapse.
Arm/Group | Main Cohort (On-treatment + Post-treatment Survival Follow-up Deaths) | Cohort 1 (On-treatment + Post-treatment Survival Follow-up Deaths)
All-Cause Mortality (participants affected / at risk) | 33/79 | 0/1
Serious Adverse Events (participants affected / at risk) | 63/79 | 0/1
Other Adverse Events (participants affected / at risk) | 79/79 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Cohort (On-treatment + Post-treatment Survival Follow-up Deaths) (N=79) | Cohort 1 (On-treatment + Post-treatment Survival Follow-up Deaths) (N=1)
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 15 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 3 | 0
Cardiac failure (Cardiac disorders) | 2 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Abdominal compartment syndrome (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 3 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 7 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Allergy to immunoglobulin therapy (Immune system disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 50 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 2 | 0
Encephalitis viral (Infections and infestations) | 2 | 0
Enterobacter infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Human herpesvirus 6 infection (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Mastoiditis (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0
Meningitis pneumococcal (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 2 | 0
Rhinovirus infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Staphylococcal abscess (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 1 | 0
Viral haemorrhagic cystitis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone giant cell tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Hypotension (Vascular disorders) | 8 | 0
Venoocclusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Cohort (On-treatment + Post-treatment Survival Follow-up Deaths) (N=79) | Cohort 1 (On-treatment + Post-treatment Survival Follow-up Deaths) (N=1)
Anaemia (Blood and lymphatic system disorders) | 25 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 5 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 13 | 0
Neutropenia (Blood and lymphatic system disorders) | 11 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 0
Tachycardia (Cardiac disorders) | 17 | 0
Abdominal pain (Gastrointestinal disorders) | 11 | 0
Constipation (Gastrointestinal disorders) | 13 | 0
Diarrhoea (Gastrointestinal disorders) | 24 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 21 | 0
Vomiting (Gastrointestinal disorders) | 25 | 0
Chills (General disorders) | 7 | 0
Face oedema (General disorders) | 8 | 0
Fatigue (General disorders) | 17 | 0
Generalised oedema (General disorders) | 5 | 0
Oedema peripheral (General disorders) | 7 | 0
Pain (General disorders) | 5 | 0
Pyrexia (General disorders) | 31 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 5 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 | 0
Cytokine release syndrome (Immune system disorders) | 37 | 0
Hypogammaglobulinaemia (Immune system disorders) | 32 | 1
Conjunctivitis (Infections and infestations) | 8 | 0
Nasopharyngitis (Infections and infestations) | 7 | 0
Rhinovirus infection (Infections and infestations) | 8 | 0
Sinusitis (Infections and infestations) | 7 | 0
Staphylococcal infection (Infections and infestations) | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 12 | 0
Activated partial thromboplastin time prolonged (Investigations) | 6 | 0
Alanine aminotransferase increased (Investigations) | 18 | 0
Aspartate aminotransferase increased (Investigations) | 18 | 0
Blood bilirubin increased (Investigations) | 12 | 0
Blood creatinine increased (Investigations) | 5 | 0
Blood fibrinogen decreased (Investigations) | 7 | 0
Blood immunoglobulin A decreased (Investigations) | 7 | 0
Blood immunoglobulin M decreased (Investigations) | 7 | 0
Blood lactate dehydrogenase increased (Investigations) | 5 | 0
C-reactive protein increased (Investigations) | 5 | 0
Electrocardiogram QT prolonged (Investigations) | 5 | 0
International normalised ratio increased (Investigations) | 9 | 0
Lymphocyte count decreased (Investigations) | 17 | 0
Neutrophil count decreased (Investigations) | 24 | 0
Platelet count decreased (Investigations) | 24 | 0
Serum ferritin increased (Investigations) | 8 | 0
White blood cell count decreased (Investigations) | 24 | 1
Decreased appetite (Metabolism and nutrition disorders) | 30 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 9 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 7 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 16 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 20 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 18 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 0
Encephalopathy (Nervous system disorders) | 7 | 0
Headache (Nervous system disorders) | 27 | 0
Somnolence (Nervous system disorders) | 5 | 0
Tremor (Nervous system disorders) | 6 | 0
Agitation (Psychiatric disorders) | 6 | 0
Anxiety (Psychiatric disorders) | 14 | 0
Confusional state (Psychiatric disorders) | 7 | 0
Delirium (Psychiatric disorders) | 7 | 0
Acute kidney injury (Renal and urinary disorders) | 9 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 16 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 0
Rash (Skin and subcutaneous tissue disorders) | 8 | 0
Hypertension (Vascular disorders) | 16 | 0
Hypotension (Vascular disorders) | 18 | 0
Coagulopathy (Blood and lymphatic system disorders) | 4 | 0
Splenomegaly (Blood and lymphatic system disorders) | 4 | 0
Adrenal insufficiency (Endocrine disorders) | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0
Pancreatitis (Gastrointestinal disorders) | 4 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 4 | 0
Immunodeficiency (Immune system disorders) | 4 | 0
Seasonal allergy (Immune system disorders) | 4 | 0
Clostridium difficile infection (Infections and infestations) | 3 | 1
Gastroenteritis (Infections and infestations) | 4 | 0
Nail infection (Infections and infestations) | 4 | 0
Oral herpes (Infections and infestations) | 4 | 0
Otitis media (Infections and infestations) | 4 | 0
Parainfluenzae virus infection (Infections and infestations) | 4 | 0
Pneumonia (Infections and infestations) | 4 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 1
Blood immunoglobulin G decreased (Investigations) | 4 | 0
Fibrin D dimer increased (Investigations) | 2 | 1
Weight increased (Investigations) | 4 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 4 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Dizziness (Nervous system disorders) | 4 | 0
Seizure (Nervous system disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 4 | 0
Dysuria (Renal and urinary disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT02435849/Prot_002.pdf
  • Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT02435849/SAP_003.pdf